CLINICAL TRIAL: NCT01025505
Title: Front-line Treatment of Ph Positive (Ph+)/Bcr-Abl Positive Acute Lymphoblastic Leukemia (ALL) With Two Tyrosine Kinase Inhibitors (TKI) (Imatinib and Nilotinib). A Phase II Exploratory Multicentric Study in Elderly Patients and in Patients Unfit for Program of Intensive Therapy and Allogeneic Stem Cell Transplantation. GIMEMA Protocol LAL1408. EudraCT 2009-01327122
Brief Title: Ph+/Bcr-Abl+ ALL Imatinib and Nilotinib Rotational Study
Acronym: LAL1408
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL1408
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Treatment; Stem Cell Transplantation
Keywords: Untreated Ph+ ALL unfit for intense therapy and allo SCT
MeSH Terms: interventions — nilotinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nilotinib — The dose of NIL is 800 mg daily (400 mg twice daily). It must be adapted according to specific guidelines in case of adverse events (AE). It cannot be increased.
Drug: Imatinib — The dose of IM is 600 mg daily (300 mg b.i.d.). It must be adapted according to specific guidelines in case of AE. It cannot be increased.

SUMMARY:
This study is an open-label, multicentric, exploratory, single arm, phase II study of adults who are either more than 60 years old, or are unfit for intensive chemotherapy and allo SCT. The patients are treated with NILOTINIB, administered orally twice daily, for 6 weeks (Course A) followed by IMATINIB, administered orally twice daily, for other 6 weeks (Course B).The courses will be repeated (rotated) for a total of 4 times or until relapse, or until it is in the interest of the patients. Prednisone (P) will be administered to all patients for 7-14 days, before TKIs, so as to make it possible to wait for the results of cytogenetic and molecular tests, and to evaluate the response to P alone, hence for another 21 days. Intrathecal therapy (IT) with MTX/AraC/DEX is mandatory, monthly, in patients without clinical-cytologic evidence of meningeal involvement, while in patients with CNS involvement it is performed twice weekly until clearance of leukemic cells, hence once weekly. IM will be administered at the dosage of 600 mg daily (300 mg twice daily) and Nilotinib at the dosage of 800 mg daily (400 mg twice daily) in all courses.

All patients are scheduled to receive at least 4 courses of either drugs, for a total of 4 courses (4 x 6 = 24 weeks). After 4 courses, patients are either allowed to continue the treatment until relapse or progression, if it is in their interest, or to discontinue the treatment and receive other therapies.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated Ph+ ALL more than 60 years old or more than 18 years old, but unfit for program of intensive therapy and allogeneic SCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | at 24 months

SECONDARY OUTCOMES:
Complete Hematological Response (CHR) rate | at 6, 12 and 24 weeks
Complete Cytogenetic Response (CCgR) rate | at 6, 12 and 24 weeks and duration of CCgR
Complete molecular response rate (CMR) | at 12 and 24 weeks and duration of CMolR
Type and number of BCR-ABL kinase domain mutations | developing during and after the study
Relationship between the response, biomarkers and gene expression profile (GEP) | At the end of study
Event-Free Survival (EFS) and Overall Survival (OS) | defined as the time from the 1st dose of corticosteroids to death or last contact
Side effects, adverse events (AE) and serious AE (SAE) | At the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Michele Baccarani, Principal Investigator — Policlinico Sant'Orsola
Locations (35):
- Italy (35):
  - Azienda Ospedaliera - Nuovo Ospedale "Torrette", Ancona
  - Dipartimento Area Medica P.O., Ascoli Piceno
  - UO Ematologia con trapianto- AOU Policlinico Consorziale di Bari, Bari
  - Ospedali Riuniti, Bergamo
  - Ist.Ematologia e Oncologia Medica L.e A. Seragnoli, Bologna
  - Sezione di Ematologia e Trapianti Spedali Civili, Brescia
  - Osp. Reg. A. Di Summa, Brindisi
  - Servizio di Ematologia - CTMO - ASL 8 P.O. Binaghi, Cagliari
  - Ospedale Ferrarotto, Catania
  - Sez.Ematologia e Dip. scienze Biomediche Arcispedale S. Anna, Ferrara
  - Clinica Ematologica - Università degli Studi, Genova
  - Ospedale Niguarda "Ca' Granda", Milan
  - Sez. di medicina Interna Oncologia ed Ematologia, Modena
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Ospedale di Rilievo Nazionale "A. Cardarelli", Napoli
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Ospedale S. Luigi Gonzaga, Orbassano
  - Università degli Studi di Padova - Ematologia ed Immunologia Clinica, Padua
  - Ospedali Riuniti 'Villa Sofia-Cervello', Palermo
  - Div. di Ematologia IRCCS Policlinico S. Matteo, Pavia
  - Div. di Ematologia di Muraglia - CTMO Ospedale San Salvatore, Pesaro
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale di Piacenza, Piacenza
  - Ospedale S.Maria delle Croci, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Rimini Ospedale "Infermi", Rimini
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - U.O. Ematologia, Azienda Ospedaliera Universitaria Senese, Siena
  - SCDO Ematologia 2 AOU S.Giovanni Battista, Torino
  - Policlinico Universitario - Clinica Ematologia, Udine
  - Policlinico G.B. Rossi, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation website — http://www.gimema.it